CLINICAL TRIAL: NCT00004875
Title: Release of TFPI by Anticoagulants in Cancer Patients by Standard or LMW Heparin
Brief Title: Heparin or Enoxaparin in Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Hau C. Kwaan MD, PhD, Northwestern University
Other Study IDs: NU 96X2; NU-96X2; NCI-G00-1670
Record Dates: First submitted 2000-03-07; First posted 2004-07-26 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Lymphoma; Thromboembolism; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; thromboembolism; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Thromboembolism; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard Heparin
  Interventions: Drug: heparin
- Enoxaprin
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: enoxaparin
  Groups: Enoxaprin
Drug: heparin
  Groups: Standard Heparin

SUMMARY:
RATIONALE: Heparin or enoxaparin may be effective in preventing the formation of blood clots in patients with cancer who are undergoing surgery to remove the tumor.

PURPOSE: Randomized clinical trial to compare the effectiveness of heparin with that of enoxaparin in patients who have cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the patterns of tissue factor pathway inhibitor (TFPI) release according to tumor type and type of anticoagulation (heparin or enoxaparin) in patients with cancer. II. Determine the incidence of portacath clots and its correlation to TFPI releasability in this patient population. III. Compare these anticoagulation drugs in terms of releasability of TFPI in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to prior chemotherapy within the past 3 weeks (yes vs no). Patients are randomized to one of two treatment arms. Arm I: Patients receive a single dose of standard heparin subcutaneously (SQ) followed by evaluation of tissue factor pathway inhibitor (TFPI) response at 5 and 10 minutes post injection. Arm II: Patients receive a single dose of enoxaparin SQ followed by evaluation of TFPI response as in arm I. Patients are followed monthly for 3 months.

PROJECTED ACCRUAL: A total of 20-200 patients will be accrued for this study over 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignancy, including lymphomas No leukemias

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Greater than 6 months Hematopoietic: Hemoglobin greater than 8.5 g/dL Platelet count greater than 100,000/mm3 No history of heparin and/or low weight molecular heparin induced thrombocytopenia No history of bleeding diathesis Hepatic: No history of coagulation factor deficiency No hepatic encephalopathy No hepatic failure No cirrhosis No hemophilia Renal: Creatinine less than 2.5 mg/dL (no greater than upper limit of normal for diabetes mellitus) Cardiovascular: No New York Heart Association class III or IV heart disease No congestive heart failure No uncontrolled hypertension (i.e., systolic blood pressure at least 180 mmHg and diastolic blood pressure at least 110 mmHg) No endocarditis No hemorrhagic stroke No prior or concurrent deep vein thrombosis Pulmonary: No prior or concurrent pulmonary embolus Other: No known allergy to enoxaparin or standard heparin No known allergy to fish (e.g., protamine sulfate) or swine products No active ulcerative disease or angiodysplasia of the gastrointestinal (GI) tract or active GI bleeding within the past 6 months No other active significant medical illness or major failure of any organ system No refusal of donor blood products secondary to religious or other reasons Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Concurrent chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: At least 1 month since prior eye, spinal cord, or CNS surgery Other: At least 1 day since prior heparin or enoxaparin At least 1 week since prior therapeutic coumadin (prior prophylactic coumadin allowed) No other concurrent anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A group of cancer patients representing a large variety of different tumor types will be observed after receiving standard heparin or enoxaprin to determine risk for thromboembolic disease.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 1996-07; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hau C. Kwaan, MD, Study Chair — Veterans Affairs Medical Center - Lakeside Chicago
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois